CLINICAL TRIAL: NCT04174248
Title: The Evaluation of Intelligence Breast Cancer Self-Management Mobile Care Application Intervention in the Quality of Life for Newly Diagnosed Non-metastatic Breast Cancer Women: Randomized Controlled Trial.
Brief Title: Breast Cancer Self-Management Mobile Care Application Intervention in the Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, I-Ching Hou, Assistant Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: YM107109E
Record Dates: First submitted 2019-11-19; First posted 2019-11-22 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Breast Cancer; Quality of Life
Keywords: breast cancer; m-Health application; self-management; life of quality
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group with BCSMS App using
  Interventions: Other: BCSMS App
- Control group (No Intervention): Control group without BCSMS App using

INTERVENTIONS:
Other: BCSMS App — Breast Cancer Using a Self-Management Support mHealth Application
  Arms: Experimental group

SUMMARY:
The aim of this study was to investigate the quality of life (QoL) for women with breast cancer in Taiwan after using the BCSMS App.

DETAILED DESCRIPTION:
After receiving their first diagnosis of breast cancer, women with stage 0 to III were randomized into intervention and control groups. Intervention group subjects used BCSMS App and the control group subjects received usual care. Two questionnaires: EORTC QLQ-C30 and EORTC QLQ-BR 23 were distributed to subjects in both arms at baseline and at 1.5 and 3 months. All evaluations were anonymous.

ELIGIBILITY:
Inclusion Criteria:

* first diagnosis of breast cancer with stage 0 to III in past year.
* aged 20 to 65 years
* had an Android/iOS smartphone;
* able to read and write in Chinese;
* willing to participate in the study and provide informed consent.

Exclusion Criteria:

* not matched to inclusion criteria
* mental illness
* serious illness and life-threatening

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2019-07-06 (Actual); Study Completion 2019-07-06 (Actual)

PRIMARY OUTCOMES:
Baseline EORTC QLQ-C30 | Baseline
  Baseline Taiwan Chinese version of the European Organisation for Research and Treatment of Cancer Quality of Life -Core 30 (version 3). The minimum and maximum values are 0 and 100, and higher scores mean a better outcome.
Change of EORTC QLQ-C30 at 1.5 month | 1.5 month
  Change from baseline Taiwan Chinese version of the European Organisation for Research and Treatment of Cancer Quality of Life -Core 30 (version 3) to 1.5 month.The minimum and maximum values are 0 and 100, and higher scores mean a better outcome.
Change of EORTC QLQ-C30 at 3 month | the 3rd month
  Change from baseline Taiwan Chinese version of the European Organisation for Research and Treatment of Cancer Quality of Life -Core 30 (version 3) to the 3rd month. The minimum and maximum values are 0 and 100, and higher scores mean a better outcome.

SECONDARY OUTCOMES:
Baseline EORTC QLQ-BR23 | Baseline
  Baseline Taiwan Chinese version of the European Organisation for Research and Treatment of Cancer Quality of Life -Breast 23 (version 3). The minimum and maximum values are 0 and 100, and higher scores mean a better outcome.
Change of EORTC QLQ-BR23 at 1.5 month | 1.5 month
  Change from baseline Taiwan Chinese version of the European Organisation for Research and Treatment of Cancer Quality of Life -Breast 23 (version 3) to 1.5 month. The minimum and maximum values are 0 and 100, and higher scores mean a better outcome.
Change of EORTC QLQ-BR23 at 3 month | the 3rd month
  Change from baseline Taiwan Chinese version of the European Organisation for Research and Treatment of Cancer Quality of Life -Breast 23 (version 3) to the 3rd month. The minimum and maximum values are 0 and 100, and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: ICing Hou, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hou IC, Lin HY, Shen SH, Chang KJ, Tai HC, Tsai AJ, Dykes PC. Quality of Life of Women After a First Diagnosis of Breast Cancer Using a Self-Management Support mHealth App in Taiwan: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Mar 4;8(3):e17084. doi: 10.2196/17084. PMID 32130181